CLINICAL TRIAL: NCT03085693
Title: Impact of Left Atrial Appendage Closure With a Closure Device on Quality of Life, Physical Capacity and Expression of Atrial Natriuretic Peptide and Brain Natriuretic
Brief Title: Impact of Left Atrial Appendage Closure on Physical Capacity.
Acronym: LAAEX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Collaborators: University of Jena (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PD Dr. med., University of Jena
Other Study IDs: SMW06
Record Dates: First submitted 2016-10-25; First posted 2017-03-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Closure of the left atrial appendage in patients with atrial fibrillation and risk for stroke is a increasing technology leading to exclusion of the left atrial appendage volume from the blood circulation and therefore protects from cardioembolic strokes- It is unclear if the volume reduction of the left atrium leads to a change in exercise capacity or Quality of life.

DETAILED DESCRIPTION:
The monocentric trial deals with the endocrinological changes as a result of closure of the left atrial appendage with a internal closure device. Specially, the changes in atrial natriuretic peptide, brain natriuretic peptide and their impact on exercise capacity is on focus of the trial. The trial is planned as a all comers trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a indication for LAA closure device Implantation

Exclusion Criteria:

* Inability to perform exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients before and after closure of the left atrial appendage
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2022-12 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
exercise capacity measured by maximal oxygen consumption | Baselina, 45 days, 6 months
  Change from baseline spiroergometry to 45 days to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, MD, PhD, Principal Investigator — University of Jena
Locations (1):
- University of Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: No